CLINICAL TRIAL: NCT02032862
Title: Multicentric, Randomized, Double Blind Study for Assessment of Efficacy and Tolerability of Sage Tablets Compared to Placebo in Menopausal Patients With Hot Flushes and Sweating
Brief Title: Efficacy and Safety of Sage Tablets Compared to Placebo in Menopausal Patients With Hot Flushes and Sweating
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient recruitment rate
Sponsor: A. Vogel AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 920157
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Menopausal Hot Flushes
Keywords: menopause, hot flushes, hot flashes, salvia, sage, sweating
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sage tablets (Experimental): Sage extract, 3400 mg , DER 1:17, in once daily application over 12 weeks treatment phase
  Interventions: Drug: Sage extract, 3400 mg , DER 1:17
- Placebo (Placebo Comparator): Placebo, matching the verum in size and appearance, in once daily application over 12 weeks treatment phase

INTERVENTIONS:
Drug: Sage extract, 3400 mg , DER 1:17
  Arms: Sage tablets

SUMMARY:
Sage tablets ( 3400 mg extract from fresh sage leaves, DER 1:17) in a once daily application over 12 treatment weeks are compared against placebo in 200 menopausal patients with ≥ 5 hot flushes daily and a Hyperhidrosis Scale score ≥ 2

ELIGIBILITY:
Inclusion Criteria:

* Menopausal since ≥ 1 year
* ≥ 5 hot flushes /24 hours
* Hyperhidrosis Scale score ≥ 2

Exclusion Criteria:

* Affections like asthma, COPD, depression, diabetes, epilepsy, hyper- and hypothyreosis, malign tumours

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Hyperhidrosis Disease Severity Scale | Week 12

SECONDARY OUTCOMES:
Change from Baseline Menopause Rating Scale / MRS | Week 12
Change from Baseline Modified Dem Tect | Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. M. Morger, Sankt Gallen, Canton of St. Gallen, Switzerland